CLINICAL TRIAL: NCT02443480
Title: Do You Have Your SPECS in Order? Development and Validation of the Saint Paul's Endoscopy Comfort Scale (SPECS) for Colonoscopy and Upper Endoscopy
Brief Title: Development and Validation of the Saint Paul's Endoscopy Comfort Scale (SPECS) for Colonoscopy and Upper Endoscopy
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Robert Enns, Dr. Robert Enns, University of British Columbia
Other Study IDs: H14-01714
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Patient Comfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators created the St. Paul's Endoscopy Comfort Score (SPECS) which includes the frequency of verbal cues, body positioning and anxiety levels with descriptions for each of the variables. Our objective is to compare the SPECS, NAPCOMs, NPAT and GS amongst different observers and to determine any correlation with patient satisfaction.

DETAILED DESCRIPTION:
Colonoscopy is used for the diagnosis and treatment of colonic lesions as well as screening and follow up of patients at risk of developing colorectal cancer. With the increasing demand for colonoscopies, the number of procedures performed in recent years has increased dramatically (Bjorkman & Popp Jr., 2006). Given that performance of a high quality colonoscopy is dependent on the expertise and technical skills of the endoscopist, quantitative and reliable methods for measurement of the quality of colonoscopy are needed. Although other colonoscopy quality indicators, such as adenoma detection rate, have been studied comprehensively (Rex, et al., 2006), patient comfort as a measure of endoscopic quality performance has not been thoroughly assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Outpatients referred to Saint Paul's Hospital for colonoscopy and upper endoscopy
* Capable of reading and understanding English

Exclusion Criteria:

* Patients who undergo colonoscopy and upper endoscopy in the same appointment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients referred to Saint Paul's Hospital for colonoscopy and upper endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Inter-observer reliability | 15-30 minutes
  To determine the inter-observer reliability for the SPECS amongst observers and the different comfort scores, NAPCOMS, GS and NPAT.
Correlation with patient's reported pain | 10-15 minutes
  To determine the correlation of SPECS, NAPCOMS, GS and NPAT with post-procedure patient reported pain and satisfaction controlling for sedation.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Bjorkman DJ, Popp JW Jr. Measuring the quality of endoscopy. Gastrointest Endosc. 2006 Apr;63(4 Suppl):S1-2. doi: 10.1016/j.gie.2006.02.022. No abstract available. PMID 16564905
- [Background] Dyson JK, Mason JM, Rutter MD. Prior hysterectomy and discomfort during colonoscopy: a retrospective cohort analysis. Endoscopy. 2014 Jun;46(6):493-8. doi: 10.1055/s-0034-1365462. Epub 2014 Apr 30. PMID 24788540
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Gelinas C, Puntillo KA, Joffe AM, Barr J. A validated approach to evaluating psychometric properties of pain assessment tools for use in nonverbal critically ill adults. Semin Respir Crit Care Med. 2013 Apr;34(2):153-68. doi: 10.1055/s-0033-1342970. Epub 2013 May 28. PMID 23716307
- [Background] Klein DG, Dumpe M, Katz E, Bena J. Pain assessment in the intensive care unit: development and psychometric testing of the nonverbal pain assessment tool. Heart Lung. 2010 Nov-Dec;39(6):521-8. doi: 10.1016/j.hrtlng.2010.05.053. PMID 20888642
- [Background] Ko HH, Zhang H, Telford JJ, Enns R. Factors influencing patient satisfaction when undergoing endoscopic procedures. Gastrointest Endosc. 2009 Apr;69(4):883-91, quiz 891.e1. doi: 10.1016/j.gie.2008.06.024. Epub 2009 Jan 18. PMID 19152911
- [Background] Kohli E, Ptak J, Smith R, Taylor E, Talbot EA, Kirkland KB. Variability in the Hawthorne effect with regard to hand hygiene performance in high- and low-performing inpatient care units. Infect Control Hosp Epidemiol. 2009 Mar;30(3):222-5. doi: 10.1086/595692. PMID 19199530
- [Background] Leonard KL. Is patient satisfaction sensitive to changes in the quality of care? An exploitation of the Hawthorne effect. J Health Econ. 2008 Mar;27(2):444-59. doi: 10.1016/j.jhealeco.2007.07.004. Epub 2007 Nov 29. PMID 18192043
- [Background] Munson GW, Van Norstrand MD, O'donnell JJ, Hammes NL, Francis DL. Intraprocedural evaluation of comfort for sedated outpatient upper endoscopy and colonoscopy: the La Crosse (WI) intra-endoscopy sedation comfort score. Gastroenterol Nurs. 2011 Jul-Aug;34(4):296-301. doi: 10.1097/SGA.0b013e3182248777. PMID 21814063
- [Background] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM. Quality indicators for colonoscopy. Gastrointest Endosc. 2006 Apr;63(4 Suppl):S16-28. doi: 10.1016/j.gie.2006.02.021. No abstract available. PMID 16564908
- [Background] Rostom A, Ross ED, Dube C, Rutter MD, Lee T, Valori R, Bridges RJ, Pontifex D, Webbink V, Rees C, Brown C, Whetter DH, Kelsey SG, Hilsden RJ. Development and validation of a nurse-assessed patient comfort score for colonoscopy. Gastrointest Endosc. 2013 Feb;77(2):255-61. doi: 10.1016/j.gie.2012.10.003. PMID 23317691
- See also: Guidelines for the Implementation of a National Quality Assurance Programme in GI Endoscopy — https://www.rcpi.ie/news/publication/guidelines-for-the-implementation-of-a-national-quality-assurance-programme-in-gi-endoscopy/